CLINICAL TRIAL: NCT02035189
Title: Observational Study Evaluating the Potential Impact of Procalcitonin Testing on Care of Stemcell Transplant Recipients and Its Performance as an Adjunct in the Diagnosis and Prognostication of Infectious Processes
Brief Title: Observational Study Evaluating the Potential Impact of Procalcitonin Testing on Care of Stemcell Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 202342
Record Dates: First submitted 2014-01-09; First posted 2014-01-14 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An observational study in evaluating the clinical impact of procalcitonin on the care of Stem cell transplant recipient and its performance as an adjunct in the diagnosis and prognostication of Infectious processes

DETAILED DESCRIPTION:
The overall goal of this project will be to provide new insights into the use of biomarkers in surveillance for infectious processes in Stem Cell Transplant recipients by evaluating the added impact of procalcitonin testing on detection of infectious processes

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-95 years with Multiple Myeloma (MM) undergoing stem cell transplantation

Exclusion Criteria:

* None

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Myeloma at UAMS receiving Stem Cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Levels of Procalcitonin | Daily up to 30 days
  Levels of Procalcitonin will be measured daily for a period not to exceed 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Senu Apewokin, MD, Principal Investigator — University of Arkansas; Naveen Sanathkumar, MD, Study Director — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States